CLINICAL TRIAL: NCT02775344
Title: Comparison of Three-dimension Versus Two-dimension Laparoscopic Ovarian Cystectomy
Brief Title: 3D Versus 2D Laparoscopic Ovarian Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Lui Man Wa, Dr, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 14-096
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Laparoscopy; ovarian cystectomy; three dimension laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- three dimension laparoscopy (Experimental): This group of patients will have laparoscopic ovarian cystectomy performed using three-dimension laparoscopy. The procedure will be performed in usual manner.
  Interventions: Device: Three dimension laparoscopy
- Two dimension laparoscopy (No Intervention): Two-dimension laparosocpy would be used in this group of patient. The procedure will be performed in usual manner.

INTERVENTIONS:
Device: Three dimension laparoscopy — Surgery will be performed either with three dimension laparoscopy or two dimension laparoscopy.
  Arms: three dimension laparoscopy

SUMMARY:
This is a prospective randomized study involving 80 patients. All participates will be given written information on 3D laparoscopy. They will be randomized according to computer-generated random sequence into two groups, 2D and 3D group. The operation will then be performed either using 2D or 3D laparoscopy. Surgeons are allowed to change to the other type of laparoscopy if difficulty encountered. After the operation, the surgeons will be required to fill in a questionnaire self-evaluating the performance using Global rating scale component of the intraoperative assessment tool (GOALS), any discomfort encountered, any need for change of laparoscopy and their preference on the type of laparoscopy.

The level of complexity of the operation, duration of operation, blood loss and complications will be recorded.

DETAILED DESCRIPTION:
Laparoscopy has greatly replaced laparotomy in most gynaecological operations including oncological procedures. Laparoscopic approach is the mainstay for ovarian cystectomy nowadays. However the loss of depth perception and dexterity remains the drawback of laparoscopy. With the development of robotic surgery, the three-dimension vision and presence of "wrist" motion allowed surgeon to perform more complicated operations in sophisticated manner. Expensive instruments and the need for prolonged time of setup restricted the extensive use of it. Having those considerations in mind, three-dimension (3D) laparoscopy is another possible alternative. With the advancement of technology in 3D vision, it may provide better precision especially in perception of depth and spatial orientation. Dizziness, nausea, headache and ocular fatique are occasional side effects in 3D surgery which created concerns of the surgeons.

There have been studies using standardized tasks shown that 3D laparoscopy will improve the performance in surgeon both objectively and subjectively especially when performing complex task. It was suggested to be able to fasten the learning curve for beginners. The operation time was shorter when laparoscopic cholecystectomy was performed using 3D imaging without any major complications encountered.

Yet evidence in the applicability and use in clinical service in gynaecological operations are still inadequate. The investigators would like to evaluate the difference of 2D versus 3D laparoscopic ovarian cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Planned for laparoscopic ovarian cystectomy
* Willing and able to participate after the study has been explained
* Those understand either Cantonese, Putonghua or English

Exclusion Criteria:

* essential data are missing from the participants records making it impossible to judge treatment outcome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Man Wa Lui, MBBS, Principal Investigator — Queen Mary Hospital, The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Storz P, Buess GF, Kunert W, Kirschniak A. 3D HD versus 2D HD: surgical task efficiency in standardised phantom tasks. Surg Endosc. 2012 May;26(5):1454-60. doi: 10.1007/s00464-011-2055-9. Epub 2011 Dec 17. PMID 22179446
- [Background] Lusch A, Bucur PL, Menhadji AD, Okhunov Z, Liss MA, Perez-Lanzac A, McDougall EM, Landman J. Evaluation of the impact of three-dimensional vision on laparoscopic performance. J Endourol. 2014 Feb;28(2):261-6. doi: 10.1089/end.2013.0344. Epub 2014 Jan 10. PMID 24059674
- [Background] Tanagho YS, Andriole GL, Paradis AG, Madison KM, Sandhu GS, Varela JE, Benway BM. 2D versus 3D visualization: impact on laparoscopic proficiency using the fundamentals of laparoscopic surgery skill set. J Laparoendosc Adv Surg Tech A. 2012 Nov;22(9):865-70. doi: 10.1089/lap.2012.0220. Epub 2012 Oct 16. PMID 23072406
- [Background] Wagner OJ, Hagen M, Kurmann A, Horgan S, Candinas D, Vorburger SA. Three-dimensional vision enhances task performance independently of the surgical method. Surg Endosc. 2012 Oct;26(10):2961-8. doi: 10.1007/s00464-012-2295-3. Epub 2012 May 12. PMID 22580874
- [Background] Cicione A, Autorino R, Breda A, De Sio M, Damiano R, Fusco F, Greco F, Carvalho-Dias E, Mota P, Nogueira C, Pinho P, Mirone V, Correia-Pinto J, Rassweiler J, Lima E. Three-dimensional vs standard laparoscopy: comparative assessment using a validated program for laparoscopic urologic skills. Urology. 2013 Dec;82(6):1444-50. doi: 10.1016/j.urology.2013.07.047. Epub 2013 Oct 2. PMID 24094658
- [Background] Vassiliou MC, Feldman LS, Andrew CG, Bergman S, Leffondre K, Stanbridge D, Fried GM. A global assessment tool for evaluation of intraoperative laparoscopic skills. Am J Surg. 2005 Jul;190(1):107-13. doi: 10.1016/j.amjsurg.2005.04.004. PMID 15972181
- [Result] Bilgen K, Ustun M, Karakahya M, Isik S, Sengul S, Cetinkunar S, Kucukpinar TH. Comparison of 3D imaging and 2D imaging for performance time of laparoscopic cholecystectomy. Surg Laparosc Endosc Percutan Tech. 2013 Apr;23(2):180-3. doi: 10.1097/SLE.0b013e3182827e17. PMID 23579515

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 women have been enrolled into the study with informed consent signed. However, their operations were rescheduled, thus did not include in the randomization.
Period: Overall Study
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy
Started | 40 | 40
Completed | 37 | 38
Not Completed | 3 | 2
Not completed — No ovarian cyst identified | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (7.0) | 36.6 (7.1) | 36.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 37 | 38 | 75
body mass index [Mean (Standard Deviation); unit: kg/m2] | 21.3 (2.6) | 23.4 (4.4) | 22.4 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: The Duration of Laparoscopic Ovarian Cystectomy
Description: The duration of laparoscopic ovarian cystectomy will be recorded. It is defined as from insertion of primary port insertion till completion of performance of ovarian cystectomy. The time required for specimen retrieval will not be included.
Time Frame: duration of operation, up to 120 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy
Number analyzed (Participants) | 37 | 38
minutes | 51.6 (36.2) | 47.6 (32.0)
Statistical Analysis 1: Comparison: Three Dimension Laparoscopy vs Two Dimension Laparoscopy; Test type: Superiority; p = 0.198, Chi-squared, Corrected; Mean Difference (Final Values) = 4

2. Primary Outcome: Global Rating Scale Component of the Intraoperative Assessment Tool (GOALS) Score
Description: Surgeons are required to fill in a questionnaire using GOALS. It involved seven aspects - depth perception, bimanual dexterity, efficiency, tissue handling, autonomy, sharpness and image resolution. Each aspects scored 0 to 5 with higher the value, better the performance. The sum of the 7 aspects were used in comparison between groups with a maximum score of 35.
Time Frame: During the operation, up to 120 minutes
Population: Chief surgeons of the operation were required to find in a questionnaire immediate postoperatively which include GOALS score assessment, any side effects experienced and their preferences for 2D/ 3D laparoscopy for the particular operation. As the assessment is on case to case basis, thus individual surgeons not recruited.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy
Number analyzed (Participants) | 37 | 38
score on a scale | 20.1 (3.3) | 20.8 (3.9)
Statistical Analysis 1: Comparison: Three Dimension Laparoscopy vs Two Dimension Laparoscopy; Test type: Superiority; p = 0.393, Chi-squared, Corrected; Mean Difference (Final Values) = 0.7

3. Secondary Outcome: Number of Surgeons Encountered Side Effects
Description: Dizziness, nausea and ocular fatique are common side effects of 3D laparoscopy. The number of surgeons experienced discomfort will be reported and any additional discomfort will be recorded.
Time Frame: during the operation, up to 120 minutes
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy
Number analyzed (Participants) | 37 | 38
Participants | 17 | 2

4. Secondary Outcome: Preference of Surgeons
Description: Surgeons need to indicate their preference of 3D or 2D laparoscopy after the surgery.
Time Frame: during the operation, up to 120 minutes
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy
Number analyzed (Participants) | 37 | 38
Participants
  Prefer 3D laparoscopy | 7 | 0
  Prefer 2D laparoscopy | 16 | 9
  No Preference | 14 | 29

5. Secondary Outcome: Need for Change of Instrument
Description: The surgeons are allowed to switch from 3D laparoscopy to tranditional 2D laparoscopy if deemed necessary by the surgeons. The reason for switch of instrument will be recorded as well.
Time Frame: during the operation, up to 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy
Number analyzed (Participants) | 37 | 38
Participants | 0 | 0

6. Secondary Outcome: Total Blood Loss During Operation
Description: The total amount of blood loss during operation was recorded.
Time Frame: during the operation, up to 120 minutes
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy
Number analyzed (Participants) | 37 | 38
ml | 58.2 (56.2) | 55.1 (64.8)

7. Secondary Outcome: Duration of Hospital Stay
Description: The total duration of hospital stay was recorded.
Time Frame: Postoperative up to 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy
Number analyzed (Participants) | 37 | 38
Days | 2.4 (1.3) | 2.6 (1.2)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Three Dimension Laparoscopy | Two Dimension Laparoscopy
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No